CLINICAL TRIAL: NCT04771780
Title: A Phase 3, Long-term, Phosphate Binder Switch Study of KHK7791 in Hyperphosphatemia Patients on Hemodialysis
Brief Title: Phosphate Binder Switch Study of KHK7791 in Hyperphosphatemia Patients on Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7791-007
Record Dates: First submitted 2021-02-16; First posted 2021-02-25 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Hyperphosphatemia
Keywords: Tenapanor; Hyperphosphatemia; Hemodialysis
MeSH Terms: conditions — Hyperphosphatemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KHK7791 (Experimental): During the dosing period, subjects administer KHK7791 twice daily just before meals.Subjects will be underwent tests at scheduled visits at least weekly until Week 12, at least once every 2 weeks after completion of Week 12 test.
  KHK7791 and phosphate binders are adjusted with the goal of controlling serum phosphorus concentration within a certain range based on the dose adjustment criteria described in the study protocol.It should be considered that phosphorus adsorbent should be switched to KHK7791 whenever feasible.
  Interventions: Drug: KHK7791

INTERVENTIONS:
Drug: KHK7791 — oral administration

SUMMARY:
To investigate the safety of repeated administration of KHK7791 for 52 weeks while switching from a phosphate-binding agent to KHK7791 in Hemodialysis patients with hyperphosphatemia.

ELIGIBILITY:
Inclusion Criteria:

1. Has voluntarily provided written informed consent to participate in the study.
2. Aged ≥ 20 years (expressed in completed years) at the time of providing informed consent.
3. Stable chronic renal failure patients who have undergone hemodialysis 3 times per week for at least 12 weeks until screening examination.
4. Dialysis conditions excluding dry weight, should have been unchanged during the last 2 weeks before screening examination.
5. The prescribed drug and dosage regimen should have been unchanged during the last 4 weeks before screening examination.
6. Serum phosphorus levels should be in the range of ≥ 3.5 and ≤ 7.0 mg/dL at screening examination.
7. If on any vitamin D, calcimimetics regimen, bisphosphonate,calcitonin preparations, selective estrogen receptor modulators or teriparatide preparations then the prescribed drug and dosage regimen should have been unchanged for the last 4 weeks before screening examination.
8. Kt/V urea ≥ 1.2 at the most recent test in routine medical practice before screening examination.

Exclusion Criteria:

1. Peritoneal dialysis was performed within 12 weeks before screening examination.
2. iPTH > 600 pg/mL (should be based on the most recent value from patient's medical records before pre-enrollment)
3. History of inflammatory bowel disease (IBD) or diarrhea predominant irritable bowel syndrome
4. History of gastrectomy or enterectomy (excluding endoscopic resection and cecectomy) or having undergone gastrointestinal tract surgery within 3 months before screening examination.
5. Subjects who used anti RANKL preparations within 6 weeks before screening examination.
6. Subjects who used anti-sclerostin antibody preparations within 12 weeks before screening examination.
7. Severe heart disease, hepatic impairment, or concurrent cirrhosis.
8. Developed cerebrovascular disease or cardiovascular disease requiring hospitalization within 6 months before screening examination.
9. Uncontrollable hypertension or diabetes
10. Subjects experienced more than 3 times diarrhea or loose stool in a day at least six BSFS score more than two days in a week.
11. Scheduled for living donor kidney transplant, change in the mode of dialysis, home hemodialysis or plans to change the dialysis center (relocate to another hospital/clinic) during the study period.
12. Any diagnosis of or treatment of malignancy within 5 years before screening examination.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-06-27 (Actual)

PRIMARY OUTCOMES:
Incidence rates of all adverse events and adverse drug reactions that occurred or worsened after the initiation of KHK7791 treatment for 52 weeks. | Dose period Week 1~52
  To investigate the safety of repeated administration of KHK7791 for 52 weeks while switching from a phosphate-binding agent to KHK7791 in Hemodialysis patients with hyperphosphatemia.

SECONDARY OUTCOMES:
Achievement of at least 30% change of the total number of daily prescription tablets of phosphorus binders and KHK7791 from baseline in the last 3 weeks of the final assessment. | Week 1~52
  To investigate the efficacy of repeated administration of KHK7791 for 52 weeks while switching from a phosphate-binding agent to KHK7791 in hyperphosphatemic subjects undergoing hemodialysis.
  Important secondary endpoint
Total daily prescription of phosphate binders and KHK7791 tablets, such as tablet counts, at each time point after the start of treatment. | Week 1~52
Achievement of at least 30% change of the total number of daily prescription tablets of phosphorus binders and KHK7791 from baseline, at each time point after the start of treatment. | Week 1~52
The change of total daily prescription of phosphate binders and KHK7791 tablets, such as tablet counts, at each time point after the start of treatment. | Week 1~52
The rate of change of total daily prescription of phosphate binders and KHK7791 tablets, such as tablet counts, at each time point after the start of treatment. | Week 1~52
Concentration of serum phosphorous levels values at each time point. | Week 1~52
Change of serum phosphorous levels from baseline values at each time point. | Week 1~52
Achievement/failure of the target serum phosphorus level (serum phosphorus level: ≤ 6.0). | Week 1~52
Time when the target serum phosphorus level (serum phosphorus level: ≤ 6.0) was achieved. | Week 1~52
Achievement/failure of the target serum phosphorus level (serum phosphorus level: ≤ 5.5). | Week 1~52
Time when the target serum phosphorus level (serum phosphorus level: ≤ 5.5) was achieved. | Week 1~52
Concentrations of such as Ca × P product levels at each time point. | Week 1~52
Changes of such as Ca × P product levels from baseline values at each time point. | Week 1~52

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Corporation Seijinkai Ikeda Hospital, Kanoya, Kagoshima-ken, Japan

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated and/or analyzed during the study sponsored by Kyowa Kirin will be available in the Vivli repository, https://vivli.org/ourmember/kyowa-kirin/ as long as conditions of data disclosure specified in the policy section of the Vivli website are satisfied.

REFERENCES:
- [Derived] Koiwa F, Sato Y, Ohara M, Nakanishi K, Fukagawa M, Akizawa T. Long-term safety and decrease of pill burden by tenapanor therapy: a phase 3 open-label study in hemodialysis patients with hyperphosphatemia. Sci Rep. 2023 Nov 4;13(1):19100. doi: 10.1038/s41598-023-45080-9. PMID 37925471